CLINICAL TRIAL: NCT02761785
Title: Gluten-free Oats and Gastrointestinal Health in Coeliac Disease, Part 2
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Kaisa Linderborg, Professor of Molecular Food Sciences (acting), University of Turku
Other Study IDs: KAURA2
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Unidentified Gastrointestinal Symptoms Following Gluten-free Oats Consumption

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal samples, urine samples and blood serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Celiacs with oat-related symptoms: Celiac patients who have self-reported gastrointestinal symptoms after ingestion of gluten-free oats
- Celiacs without oat-related symptoms: Celiac patients who include gluten-free oats in their diet and have no symptoms related to oats
- Healthy controls: Healthy controls (without celiac disease) who include oats in their diet
- Non-celiac gluten sensitive subjects: Subjects with manifestations precipitated by ingestion of gluten in whom celiac disease and wheat allergy are excluded.

SUMMARY:
The research aims to investigate the effects of gluten-free oats to the gastrointestinal health in celiac disease patients and healthy subjects. The effects of gluten-free oats on the several intestinal parameters, on the composition of the gut microbiota as well as on the metabolic profile of celiac patients and healthy controls will be studied. The study is divided into two parts.

Part 1 will be conducted as a double-blind, randomized and placebo-controlled cross-over study. Healthy subjects will be recruited to the study. The aim is to recruit 15 participants for the part 1. The study will be conducted with a cross-over setting, where the subjects will go through exposure meals and SmartPill ingestion three times (two different oat products and placebo) in a randomized order. The study meals are identical in appearance and fiber content. After consuming the meal subjects will ingest the SmartPill capsule, which will send data on intestinal pH, pressure and temperature to the external portable device. Before and during the passage of capsule the subjects will fill a symptom and food diary. The capsule will exit the body in 1 to 3 days and the data collected by the external device will be collected and analyzed. Before the oat/placebo exposure the subjects will give a fecal and a blood sample. In addition, 36 hours urine samples will be collected.

In part 2 celiac disease patients, non-celiac gluten sensitive subjects and healthy controls will be recruited and they will be divided into four groups: oat-avoiding celiacs (1), oat-consuming celiacs (2), non-celiac gluten sensitive subjects (3) and healthy controls (4). Recruiting aim for each group is 15 subjects. In addition to dietary data, a blood, and a fecal sample will be collected from the subjects. The gut microbiota will be analyzed from the fecal samples. The metabolic products will be analyzed from the fecal, urine and blood samples. The gut microbiota composition will be analyzed with next-generation DNA sequencing techniques.

ELIGIBILITY:
Inclusion Criteria:

* Celiac disease diagnosed with duodenal biopsy (only celiac groups)
* In remission and maintained gluten-free diet >1 year (only celiac groups)
* Usage of oats in their diet (only oat-using celiacs and healthy controls)
* BMI 18,5 - 30
* Normal liver, thyroid and kidney functions

Exclusion Criteria:

* Medication that majorly affects GI tract (e.g. laxatives, antacids)
* Antibiotic treatment within the last 6 months
* Blood donation or participating in another clinical trial within the last month

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group 1:Celiac patients who have self-reported gastrointestinal symptoms after ingestion of gluten-free oats
  Group 2: Celiac patients who include gluten-free oats in their diet and have no symptoms related to oats
  Group 3: Non-celiac gluten sensitive subjects
  Group 4: Healthy controls (without celiac disease) who include oats in their diet
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota composition | Measured from single time point sampling
  Fecal microbiota diversity and composition analyzed from fecal sample
Metabolic status | Measured from single time point sampling
  Metabolic status analyzed by the amount of metabolic products found in fecal, urine and serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Linderborg, PhD, Principal Investigator — Associate professor
Locations (1):
- Department of Biochemistry, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided